CLINICAL TRIAL: NCT04127838
Title: Low Vision Occupational Therapy in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Marissa Dean, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-300003853
Record Dates: First submitted 2019-10-10; First posted 2019-10-16 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Occupational Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low Vision Occupational Therapy (Experimental): The anticipated low vision occupational therapy intervention strategy includes training participants to compensate for their vision more effectively for increased participation in ADLs and IADLs.
  Interventions: Behavioral: Low Vision Occupational Therapy

INTERVENTIONS:
Behavioral: Low Vision Occupational Therapy — Occupational therapy may include methods to effectively modify environments (such as addition of task lighting), training in the use of assistive technology (such as voice activated devices), teaching new skills (such as sensory substitution) and prevention of accidents and injury (such as home safety modifications).
  Other Names: Occupational Therapy

SUMMARY:
The primary aim of this study is to determine whether low-vision occupational therapy improves quality of life in Parkinson's Disease (PD) patients. Low-vision occupational therapy has not been previously studied in PD patients, and we suspect that this is a beneficial treatment option for PD patients as vision impairment is common in the PD patient population. Our primary objective will assess whether quality of life was improved following a low-vision occupational therapy session.

DETAILED DESCRIPTION:
This project will be an exploratory study that will evaluate the benefits of low vision occupational therapy in the treatment of PD using the Revised Self-Report Assessment of Functional Visual Performance (R-SRAFVP) as the primary outcome measure. This tool assesses 33 vision-dependent ADLs ranging from personal care, leisurely activities, clothing management, meal preparation, etc. Patients are able to rank their ability to complete these tasks as independent, minimally difficult, moderately difficult, greatly difficult, unable, or not applicable. This will allow us to capture potential changes in the patient's ability to complete vision-specific ADLs following low vision occupational therapy. In addition, we will also evaluate quality of life using the Parkinson's Disease Questionnaire (PDQ-39), to compare this broad outcome measure with the R-SRAFVP.

ELIGIBILITY:
Inclusion Criteria:

* 18 and older
* seen at UAB Movement Disorders Clinic
* diagnosis of idiopathic Parkinson's Disease
* able to read, speak, and understand spoken English.

Exclusion Criteria:

* minors
* cognitively impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
Change in Activities of Daily Living | Changes measured in the R-SRAFVP from the initial visit as compared to the visit six months later.
  Revised Self-Report Assessment of Functional Visual Performance (R-SRAFVP). This tool assesses 33 vision-dependent ADLs ranging from personal care, leisurely activities, clothing management, meal preparation, etc. Patients are able to rank their ability to complete these tasks as independent, minimally difficult, moderately difficult, greatly difficult, unable, or not applicable.

SECONDARY OUTCOMES:
Change in quality of life | Changes measured in the PDQ-39 from the initial visit as compared to the visit six months later.
  Parkinson's Disease Questionnaire (PDQ-39); The PDQ-39 assesses how often people affected by Parkinson's experience difficulties across 8 dimensions of daily living including relationships, social situations and communication

CONTACTS AND LOCATIONS:
Overall Officials: Marissa Dean, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No